CLINICAL TRIAL: NCT02420899
Title: Effect of Different Doses of Rosuvastatin Therapy on Regression of Critical Coronary Atherosclerosis in Chinese ACS Patients
Brief Title: Different Doses of Rosuvastatin Therapy on Regression of Critical Coronary Atherosclerosis in ACS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hui Chen, Hui Chen,Director,Clinical Professor,Principal Investigator, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 40068860-9
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome
Keywords: IVUS; ACS
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Statins,lipid-lowering drugs (Experimental): rosuvastatin 10mg or 20mg per day，pro
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — 10mg/d or 20mg/d,po
  Other Names: crestor

SUMMARY:
The purpose of this study is to determine whether Rosuvastatin 10mg/d or 20mg/d for 36 weeks can regress critical coronary atherosclerosis as determined by IVUS imaging in Chinese Acute Coronary Syndrome (ACS) patients.

DETAILED DESCRIPTION:
This is a prospective, open-label, parallel group study to evaluate the efficacy of rosuvastatin 10mg/d or 20mg/d on critical coronary atherosclerosis in Chinese ACS patients. The anticipated duration of the study is approximately 36 weeks, Patients with angiographic luminal diameter narrowing in any non-culprit site between 40%-70% will be enrolled from the study site. The primary efficacy parameter is the percent change of Total Atheroma Volume (TAV) of critical coronary atherosclerosis after 36 weeks of treatment.

For inclusion in the study subjects should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. 18 to 75 years old ACS patients, male or female
3. The angiographic luminal diameter narrowing in any non-culprit site is between 40%-70%
4. statin-naive, defined as receiving no statin therapy within 3 monthsThe primary efficacy variable of the study is percent change of TAV from baseline after rosuvastatin 10mg/d or 20mg/d for 36 weeks as determined by IVUS imaging.

The secondary efficacy variables are:

* Change of blood lipid level from baseline at 12th, 24th, 36nd week
* Change of inflammatory markers from baseline at 36nd week
* Change of Percent Atheroma Volume (PAV) as determined by IVUS imaging at 36nd week

ELIGIBILITY:
Inclusion Criteria:

1.Provision of informed consent prior to any study specific procedures; 2.18 to 75 years old ACS patients, male or female; 3.The angiographic luminal diameter narrowing in any non-culprit site is between 40%-70%; 4.statin-naive, defined as receiving no statin therapy within 3 months;

Exclusion Criteria:

1. Have received statin therapy within 3 months;
2. The angiographic luminal diameter narrowing in any coronary vessels is more than 70%;
3. Active liver disease, ALT≥3*ULN;
4. Renal function damage, CrCl<30ml/min;
5. Myopathy;
6. Pregnancy, lactation female;
7. Using cyclosporine;
8. Patients with uncontrolled triglyceride levels TG≥5.65 mmol／L;
9. Poorly controlled diabetes (HbA1c≥10%）Hypersensitivity to rosuvastatin or any of the recipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Percent Atheroma Volume (PAV) | 36 weeks
  Percent Atheroma Volume

SECONDARY OUTCOMES:
inflammatory marker levels | 36 weeks
  MCP-1, VCAM-1 level and mRNA level of ICAM-1, CCR2

OTHER OUTCOMES:
Total Atheroma Volume (TAV) | 36 weeks
  Total Atheroma Volume
lipid level | 36 weeks
  LDL-C,HDL-C,TC,TG
safety and tolerability as assessed by blood biochemistry, blood routines and urine routines | 36 weeks
  blood biochemistry, blood routines and urine routines

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Liu Qingbo, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] 1.Liao J K, Laufs U. Pleiotropic effects of statins[J]. Annual review of pharmacology and toxicology, 2005, 45: 89. 2.Davignon J. Beneficial cardiovascular pleiotropic effects of statins[J]. Circulation, 2004, 109(23 suppl 1): III-39-III-43. 3.Falk E, Shah P K, Fuster V. Coronary plaque disruption[J]. Circulation, 1995, 92(3): 657-671. 4. Nissen SE, Nicholls SJ, Sipahi I, et al.Effect of very high-intensity statin therapy on regression of coronary atherosclerosis:the ASTEROID trial. JAMA, 2006; 295: 1556-65. 5. Lee CW, et al. Comparison of Effects of Atorvastatin(20mg) Versus Rosuvastatin(10mg) Therapy on Mild Coronary Atherosclerosis Plaques(from the ARTMAP Trial).Am J Cardiol, 2012; 109:1700-1704.